CLINICAL TRIAL: NCT04615949
Title: Study to Evaluate the Efficacy and Safety of CardiolRx™ in Patients With COVID-19 and Cardiovascular Disease or Risk Factors A Double-blind, Placebo-controlled Trial
Brief Title: Cannabidiol in Patients With COVID-19 and Cardiovascular Disease or Risk Factors
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The changing nature of COVID-19 including a more vaccinated population, increasing natural population immunity, milder variants and other related factors has meant that it is no longer realistic to recruit the patients in a reasonable time frame.
Sponsor: Cardiol Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CARDIOL 100-03
Record Dates: First submitted 2020-11-02; First posted 2020-11-04 (Actual); Results first posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2022-10

CONDITIONS: COVID-19; Cardiovascular Diseases; Cardiovascular Risk Factor
MeSH Terms: conditions — COVID-19; Cardiovascular Diseases | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, parallel study, randomization 1:1
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cannabidiol, pharmaceutically produced with < 5 ppm THC (Experimental): CardiolRx
  Interventions: Drug: Cannabidiol, pharmaceutically produced with < 5 ppm THC
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol, pharmaceutically produced with < 5 ppm THC — CardiolRx 2.5 mg/kg to 7.5 mg/kg of body weight b.i.d taken orally with food
  Other Names: CardiolRx
  Arms: Cannabidiol, pharmaceutically produced with < 5 ppm THC
Drug: Placebo — Placebo 2.5 mg/kg to 7.5 mg/kg of body weight b.i.d taken orally with food
  Arms: Placebo

SUMMARY:
Non-critical patients, hospitalized within the previous 24 hours who tested positive for COVID-19 and have a prior history of cardiovascular disease (CVD) and/or significant risk factors for CVD will be treated for 28 days.

DETAILED DESCRIPTION:
Multi-center, double-blind, randomized, placebo-controlled, parallel group design. 1:1 randomization.

Screening (Day 0-1): Patients hospitalized for COVID-19 within the past 24 hours will be screened. If patient consent can be obtained, baseline assessments will be carried out: Physical examination (including vital signs), ECG including QTc interval assessment, echocardiogram to measure left-ventricular ejection fraction (LVEF), chest X-ray, local laboratory (including CBC, AST/ALT, alkaline phosphatase, bilirubin, creatinine/eGFR, INR, pregnancy test (in women with child-bearing potential only), lymphocyte count and LDH. A C-SSRS will also be completed. Frozen plasma will be retained for central analysis of CardiolRx™ levels, hs-troponin, NT-proBNP, D-dimer as well as inflammatory markers (hs-CRP, ferritin, TNF-alpha, IL-1 beta, IL-6, IL-10).

If all eligibility criteria are met, the patient will be randomized to either CardiolRx™ or placebo.

Study treatment will be initiated immediately after all baseline assessments have been completed and the patient is randomized (Day1). Oral administration is as follows:

* Day 1 and Day 2: Initial dose: 2.5 mg/kg of body weight b.i.d. with food: CardiolRx™ or placebo
* Day 3 and Day 4: Increased to 5 mg/kg of body weight b.i.d. with food: CardiolRx™ or placebo
* Day 5 to Day 28: Increased to 7.5 mg/kg of body weight b.i.d. with food: CardiolRx™ or placebo For the first 7 days and on Day 10, an ECG will be recorded 4 hours post morning dose with QTc intervals measured. If the QTc interval is >500 msec or an increase of > 60 msec from baseline is observed, the study medication must be stopped immediately.

If the next higher dose is not tolerated for other reasons, the dose will be reduced to the previous tolerated dose. The highest tolerated dose will be administered until Day 28.

If the patient is discharged before Day 10, the assessments up to Day 10 will be carried out as home visits. After Day 10, all remaining scheduled assessments will be carried out during out-patient visits (or home visits, if out-patient visits are not feasible).

In addition to prolongation of the QTc intervals, careful observation is required to detect other Adverse Drug Reactions (ADRs) and Drug-Drug Interactions (DDIs). Because CardiolRx™, may inhibit the metabolism of other drugs, new symptoms may represent toxicity from a concomitant medication that had previously been well tolerated.

A nasopharyngeal swab will also be done every day until Day 7 and on Day 14 to test for presence of the SARS-CoV-2 virus.

After Day 7, assessments will be carried out on a weekly basis except for as noted above on Day 10.

Frozen plasma will be retained for central analysis of CardiolRx™ levels, hs-troponin, NT-proBNP, D-dimer, inflammatory markers (hs-CRP, ferritin, TNF-alpha, IL-1 beta, IL-6, IL-10) and additional parameters of interest every two days until Day 7 as well as on day 28.

The assessments on Day 28 include the following: Physical examination (including vital signs), ECG (recorded 4 hours post morning dose for measurement of QTc interval), echocardiogram to measure LVEF, chest X-ray, local laboratory assessments, including CBC, AST/ALT, alkaline phosphatase, bilirubin, creatinine/eGFR, INR, lymphocyte count and LDH. In addition, a C-SSRS will be completed and the patient will be asked to answer a PICQ.

Further follow-up visits are scheduled for Day 45 and Day 60 post randomization. These include a clinical assessment (including vital signs) as well as the completion of the PICQ (PICQ on Day 60 only). Any changes in concomitant medications and (S)AEs will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 years of age or older 2. Hospitalized for COVID-19 with the most recent test positive*; not receiving or likely to receive invasive mechanical ventilation within the next 24 hours 3. Prior history of at least one of: i) CVD [cardiovascular (CV), cerebrovascular or peripheral vascular diagnoses], ii) Age > 64, iii) Diabetes (DM), iv) Hypertension (HTN), v) Abnormal serum lipids, vi) Obesity (BMI > or equal 30 or waist circumference >102 cm [40"] for men and >88 cm [35"] for women), vii) Current smoker

* Must be PCR test.

Exclusion Criteria:

1. Patients who have received vasopressors, extracorporeal membrane oxygenation and mechanical ventilation within last 30 days
2. Background of cardiac transplant surgery
3. Implanted defibrillator (ICD) in the last three months
4. Implanted left-ventricular assist device (LVAD)
5. Acute coronary syndrome (ACS) within 30 days
6. Percutaneous coronary intervention (PCI) within 30 days
7. Receiving any immuno-suppressive agent other than dexamethasone
8. History of QTc interval prolongation
9. QTc interval > 500 msec
10. Treated with strong inducers of CYP3A4 or CYP2C19
11. Chronic renal failure, determined as eGFR < 30 ml/min
12. Elevated alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 times the upper limit of normal (ULN) or ALT or AST >3x ULN plus bilirubin >2x ULN
13. Bacterial sepsis, defined as documented bacteremia at the time of presentation or other active bacterial infection
14. Current participation in any research study involving investigational drugs or devices with the exception of dexamethasone, remdesivir, baricitinib plus remdesivir, convalescent plasma or monoclonal antibodies against the SARS-CoV-2 virus or any other therapy approved under emergency use in the region for treatment of COVID-19
15. Inability or unwillingness to give informed consent
16. Ongoing drug, alcohol or cannabis abuse
17. Women who are pregnant or breastfeeding
18. Any factor, which would make it unlikely that the patient can comply with the study procedures
19. Hemoglobin <8.5 gm/dL
20. Leukocyte count < 3000/ mm3
21. Platelets < 100,000 / mm3
22. Current diagnosis of cancer, with the exception of non-melanoma skin cancer
23. Showing suicidal tendency as per the Columbia-Suicide Severity Rating Scale (C-SSRS) administered at screening
24. Any cannabinoid intake in the past month
25. Body weight > 170 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis McNamara, MD, Study Chair — University of Pittsburgh
Locations (20):
- United States (7):
  - Valleywise Health Medical Center, Phoenix, Arizona
  - JY Research Institute, Cutler Bay, Florida
  - Westchester General Hospital, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - University of Texas Health Science Center, San Antonio, Texas
  - Baylor Scott & White Health - Temple, Temple, Texas
- Brazil (12):
  - Science Valley Research Institute, Campo Largo, Paraná
  - Universidade Estadual de Maringa, Maringá, Paraná
  - Hospital São Lucas PUCRS, Porto Alegre, Rio Grande do Sul
  - Irmandade Santa Casa de Misericórdia, Porto Alegre, Rio Grande do Sul
  - Núcleo de Ensino e Pesquisa do Instituto Mário Penna, Conjunto ACM, Santa Maria
  - Fundação Pio XII - Hospital de Amor Barretos, Barretos, São Paulo
  - IPECC-Instituto de Pesquisa Clínica de Campinas, Campinas, São Paulo
  - Instituto do Coração do HCFMUSP, Cerqueira César, São Paulo
  - SVRI- Irmandade de Santa Casa de Misercordia de Santos, Jabaquara, São Paulo
  - Science Valley Research Institute, Santo André, São Paulo
  - Fundação Faculdade Regional de Medicine de Sao Jose do Rio Preto (SJRP), São José do Rio Preto, São Paulo
  - Complexo Hospitalar de Niteroi- Centro de Pesquisa Clinica, Rio de Janeiro
- TecSalud, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Yes
The data will become available once the study has been published
Supporting Information: Study Protocol
Time Frame: Data will become available in Q4 2022
Access Criteria: Access to the journal in which article has been published

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cannabidiol, Pharmaceutically Produced With < 5 Ppm THC | Placebo
Started | 45 | 45
Completed | 41 | 37
Not Completed | 4 | 8
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Lost to Follow-up | 2 | 2
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cannabidiol, Pharmaceutically Produced With < 5 Ppm THC | Placebo | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (14.86) | 62.0 (12.95) | 61.2 (13.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 26 | 25 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 42 | 84
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 28 | 27 | 55
  More than one race | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 26 | 51
  Brazil | 6 | 4 | 10
  Mexico | 14 | 15 | 29
Obesity [Count of Participants; unit: Participants] | 19 | 23 | 42
Diabetes [Count of Participants; unit: Participants] | 17 | 19 | 36
Hyperlipidemia [Count of Participants; unit: Participants] | 7 | 9 | 16
Hypertension [Count of Participants; unit: Participants] | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality
Description: Proportions of patients not surviving
Time Frame: 28 days post randomization
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Cannabidiol, Pharmaceutically Produced With < 5 Ppm THC | Placebo
Number analyzed (Participants) | 45 | 45
Participants | 0 | 2

ADVERSE EVENTS:
Time Frame: 60 days
Arm/Group | Cannabidiol, Pharmaceutically Produced With < 5 Ppm THC | Placebo
All-Cause Mortality (participants affected / at risk) | 0/45 | 2/44
Serious Adverse Events (participants affected / at risk) | 5/45 | 4/44
Other Adverse Events (participants affected / at risk) | 24/45 | 23/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cannabidiol, Pharmaceutically Produced With < 5 Ppm THC (N=45) | Placebo (N=44)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1)
ALT increase (Investigations) | 0 (0) | 1 (1)
QTC segment prolongation (Investigations) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cannabidiol, Pharmaceutically Produced With < 5 Ppm THC (N=45) | Placebo (N=44)
Nausea (Gastrointestinal disorders) | 5 | 2
Constipation (Gastrointestinal disorders) | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 3
Headache (Nervous system disorders) | 4 | 3
Dysgeusia (Nervous system disorders) | 3 | 2
Dizziness (Nervous system disorders) | 0 | 3
Tachycardia (Cardiac disorders) | 0 | 3
Hypertension (Vascular disorders) | 3 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 2
Taste disorder (Nervous system disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute respiratory distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Left ventricular hypertrophy (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Fungal infection (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Blood glucose increased (Infections and infestations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Electrocardiogram QT increased (Investigations) | 1 | 0
Oedema peripheral (General disorders) | 2 | 1
Chest discomfort (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Secretion discharge (General disorders) | 1 | 0
Insomnia (Investigations) | 2 | 2
Nightmare (General disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 0
Renal impairement (Renal and urinary disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-09-23): https://cdn.clinicaltrials.gov/large-docs/49/NCT04615949/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT04615949/SAP_001.pdf